CLINICAL TRIAL: NCT05621967
Title: Phonation Therapy to Improve Symptoms and Lung Physiology in Patients Referred for Pulmonary Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in location of Pulmonary Rehab at our institution
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Vidya Krishnan, Professor of Medicine: Pulmonary, Critical Care and Sleep Medicine, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000152
Record Dates: First submitted 2022-09-16; First posted 2022-11-18 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized control trial. Randomization for each subject occurs twice. First: One of two types of intervention. Second: Sequence for intervention and normal breathing sessions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Silent Breathing / Tonation Breathing Techniques (TBT) (Experimental): Twice a week during the patient's 8 weeks of pulmonary rehabilitation:
  1. For first 4 weeks, twice a week - 20 min of silent quiet breathing while sitting.
  2. Next 4 weeks, twice a week - 20 min of TBT guided by a facilitator virtually
  Interventions: Behavioral: Tonation Breathing Techniques; Behavioral: Silent Breathing
- Silent Breathing / Music Driven Vocal Exercises (MDVE) (Experimental): Twice a week during the patient's 8 weeks of pulmonary rehabilitation:
  1. For first 4 weeks, twice a week - 20 min of silent quiet breathing while sitting.
  2. Next 4 weeks, twice a week - 20 min of MDVE guided by a facilitator in-person
  Interventions: Behavioral: Music Driven Vocal Exercises; Behavioral: Silent Breathing
- Tonation Breathing Techniques (TBT) / Silent Breathing (Experimental): Twice a week during the patient's 8 weeks of pulmonary rehabilitation:
  1. For first 4 weeks, twice a week - 20 min of TBT guided by a facilitator virtually
  2. Next 4 weeks, twice a week - 20 min of silent quiet breathing while sitting.
  Interventions: Behavioral: Tonation Breathing Techniques; Behavioral: Silent Breathing
- Music Driven Vocal Exercises (MDVE) / Silent Breathing (Experimental): Twice a week during the patient's 8 weeks of pulmonary rehabilitation:
  1. For first 4 weeks, twice a week - 20 min of MDVE guided by a facilitator in-person
  2. Next 4 weeks, twice a week - 20 min of silent quiet breathing while sitting.
  Interventions: Behavioral: Music Driven Vocal Exercises; Behavioral: Silent Breathing

INTERVENTIONS:
Behavioral: Tonation Breathing Techniques — Tonation and Breathing Techniques (TBT): consist of a combination of organic inhalation and controlled exhalation with tonation. This will be guided by a trained facilitator, and the entire exercise will take 20 minutes. This will include guided relaxed breathing, mindful breathing, patterned tonation, nasal tonation, and pursed lip tonation.
  Other Names: TBT
  Arms: Silent Breathing / Tonation Breathing Techniques (TBT); Tonation Breathing Techniques (TBT) / Silent Breathing
Behavioral: Music Driven Vocal Exercises — Music Driven Vocal Exercises (MDVE): A Music Therapy procedure will be implemented by a trained facilitator, utilizing an accompanying instrument (ie, guitar or Autoharp) and moving stepwise up and down within a scale of 8 whole steps. The total length of the procedure is 20-25 minutes. This will include vocal exercises, and melodic exercises alternating with speaking,
  Other Names: MDVE
  Arms: Music Driven Vocal Exercises (MDVE) / Silent Breathing; Silent Breathing / Music Driven Vocal Exercises (MDVE)
Behavioral: Silent Breathing — Patient will sit in a quiet room and focus on silent breathing x 20 min.

SUMMARY:
To investigate Phonation therapy to improve symptoms and lung physiology in patients referred for pulmonary rehabilitation. The study design will be a randomized controlled trial. The primary outcome is improvement in patient symptoms (Borg dyspnea score). Secondary outcomes are improvement in time of breath hold, forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), negative inspiratory force (NIF) and improvement in quality of life. The investigators will be investigating tonation breathing techniques (TBT) exercises and music-driven vocal exercises (MDVE). The study population would be patients who are referred to pulmonary rehabilitation (PR) for symptomatic chronic lung disease. The calculated sample size for the study would be 16 patients and the duration of the study would be 8 weeks. The study would be performed after the participant's pulmonary rehabilitation session.

DETAILED DESCRIPTION:
Patients who are referred for pulmonary rehabilitation for chronic lung disease and/or post-COVID19 therapy, and who have had pulmonary function testing already will be approached. Pulmonary rehabilitation is an 8-week program (meeting 3 times per week for the 8 weeks). Pulmonary rehabilitation (PR) is the standard of care for patients with chronic lung diseases and or post-COVID-19 therapy. Eligible study participants will be called prior to their introductory PR session to explain the research project, and those who are interested will be given full information and offered time to ask questions. The investigators find this necessary for logistics, given many of the PR patients rely on scheduled transportation to/from PR and this will allow those who are interested in obtaining more information and to consent to the study to arrange for appropriate transportation. Informed consent will be done in person on an individual basis at their introductory PR session, with 1:1 discussion with the study staff and the patient.

As this is a pilot study to determine feasibility, and preliminary data (as no data are currently available for this patient population), the investigators propose 16 participants in total, 4 in each arm of the study. Randomization will occur by random number generator (1-4 for each arm proposed).

Once informed consent is obtained, patients will be randomized to 4 arms of the study. Randomization will be performed using a random number generator.

1. Comparing tonation breathing technique (TBT) to normal breathing:

   1. Of the 8 weeks of PR, first 4 weeks will be sessions of normal breathing exercises for 20 minutes, then subsequent 4 weeks will be with TBT intervention for 20 minutes.
   2. Of the 8 weeks of PR, the first 4 weeks will be with TBT intervention for 20 minutes, then the next 4 weeks will be of sessions of normal breathing exercises for 20 minutes.
2. Comparing MDVE to normal breathing:

   1. Of the 8 weeks of PR, the first 4 weeks will be sessions of normal breathing exercises for 20 minutes, then the subsequent 4 weeks will be with Music Driven Vocal Exercises (MDVE) intervention for 20 minutes.
   2. Of the 8 weeks of PR, the first 4 weeks will be with MDVE intervention for 20 minutes, then the next 4 weeks will be of sessions of normal breathing exercises for 20 minutes.

These interventions would be performed after the usual PR time when patients would be normally discharged home. Therefore, no additional monitoring is expected.

Pulmonary function testing is standard for all patients who receive PR - testing before and after PR is routine clinical course. The investigators propose an additional pulmonary function test (PFT) study at 4 weeks, as part of the research protocol (covered by the Department of Medicine funding)

In summary, the interventions for research purposes will include:

1. 20-minute sessions after PR for intervention (TBT or MDVE) or normal breathing for twice a week for the 8 weeks they are participating in PR.
2. PFT at end of week 4

Proposed subjective outcomes are routinely asked of PR patients, but will be collected at baseline, at 4 weeks (mid-way), and at 8 weeks (end) of PR. Proposed objective outcomes:

1. For FEV1, FVC - these are routinely collected at baseline and at end of PR. The investigators propose an additional PFT study at 4 weeks, covered by the DOM Faculty Development Fund.
2. For peak flow and NIF - these are procedures that ask for patients to breathe maximally for inspiration and expiration. They are not routine measures collected but are routine bedside measurements for pulmonary patients that can be collected for any person without any additional risk or cost.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* English-speaking and reading patient
* Able to consent for study
* Referred for pulmonary rehabilitation for chronic lung disease (including long COVID19 syndrome, COPD, ILD, PH)
* Baseline Borg dyspnea score as moderate (score 3) or higher.
* Has baseline pulmonary function testing available in electronic medical record.

Exclusion Criteria:

• Cannot commit to staying an extra 30 min after Pulmonary Rehabilitation sessions for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Borg dyspnea score | 8 weeks
  subjective score of dyspnea

SECONDARY OUTCOMES:
FEV1 | 4 and 8 weeks
  forced expiratory volume in 1 second
Borg dyspnea score | 4 weeks
  subjective score of dyspnea
Breath hold | 4 weeks, 8 weeks
  time in seconds participant can hold breath
quality of life (QOL) | 4 weeks, 8 weeks
  questionnaire on quality of life
forced vital capacity (FVC) | 4 weeks, 8 weeks
  forced vital capacity
peak flow | 4 weeks, 8 weeks
  peak flow
negative inspiratory force (NIF) | 4 weeks, 8 weeks
  negative inspiratory force

CONTACTS AND LOCATIONS:
Overall Officials: Vidya Krishnan, MD, MHS, Principal Investigator — Case Western Reserve University, MetroHealth Campus
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostermann T, Schmid W. Music therapy in the treatment of multiple sclerosis: a comprehensive literature review. Expert Rev Neurother. 2006 Apr;6(4):469-77. doi: 10.1586/14737175.6.4.469. PMID 16623646
- [Background] Garcia-Casares N, Martin-Colom JE, Garcia-Arnes JA. Music Therapy in Parkinson's Disease. J Am Med Dir Assoc. 2018 Dec;19(12):1054-1062. doi: 10.1016/j.jamda.2018.09.025. PMID 30471799
- [Background] Canga B, Azoulay R, Raskin J, Loewy J. AIR: Advances in Respiration - Music therapy in the treatment of chronic pulmonary disease. Respir Med. 2015 Dec;109(12):1532-9. doi: 10.1016/j.rmed.2015.10.001. Epub 2015 Oct 19. PMID 26522499
- [Background] Mathis DR. Melodic sculpturing: the art and science of singing. Bloomington, IN: AuthorHouse, 2009
- [Background] Price, Kate. The effects of vocal function exercises on the lung function of trained female singers: a pilot investigation. Diss. Victoria University, 2003.
- [Background] McNamara RJ, Epsley C, Coren E, McKeough ZJ. Singing for adults with chronic obstructive pulmonary disease (COPD). Cochrane Database Syst Rev. 2017 Dec 19;12(12):CD012296. doi: 10.1002/14651858.CD012296.pub2. PMID 29253921
- [Background] DRAPER MH, LADEFOGED P, WHITTERIDGE D. Respiratory muscles in speech. J Speech Hear Res. 1959 Mar;2(1):16-27. doi: 10.1044/jshr.0201.16. No abstract available. PMID 13655288
- [Background] Bouhuys A, Proctor DF, Mead J. Kinetic aspects of singing. J Appl Physiol. 1966 Mar;21(2):483-96. doi: 10.1152/jappl.1966.21.2.483. No abstract available. PMID 5934452
- [Background] Leanderson, R.; Sundberg, J. (1988). Breathing for singing. , 2(1), 2-12. doi:10.1016/S0892-1997(88)80051-1
- [Background] Leanderson R, Sundberg J, von Euler C. Role of diaphragmatic activity during singing: a study of transdiaphragmatic pressures. J Appl Physiol (1985). 1987 Jan;62(1):259-70. doi: 10.1152/jappl.1987.62.1.259. PMID 3558185
- [Background] Huang J, Yuan X, Zhang N, Qiu H, Chen X. Music Therapy in Adults With COPD. Respir Care. 2021 Mar;66(3):501-509. doi: 10.4187/respcare.07489. Epub 2020 Nov 3. PMID 33144384
- [Background] Sliwka A, Nowobilski R, Polczyk R, Nizankowska-Mogilnicka E, Szczeklik A. Mild asthmatics benefit from music therapy. J Asthma. 2012 May;49(4):401-8. doi: 10.3109/02770903.2012.663031. Epub 2012 Mar 7. PMID 22397390
- [Background] Morrison, Ian, and S. M. Clift.

DOCUMENTS (1):
  • Study Protocol (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT05621967/Prot_000.pdf